CLINICAL TRIAL: NCT05034250
Title: Iron Status in Women With Infertility and Controls - a Prospective Case-control Study
Brief Title: Iron Status in Female Infertility and Recurrent Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Vifor Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Johannes Ott, Associate Professor, Consultant Physician, Medical University of Vienna
Other Study IDs: 20210608
Record Dates: First submitted 2021-07-19; First posted 2021-09-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Miscarriage; Infertility; Iron-deficiency
Keywords: Iron status; Recurrent Miscarriage; Infertility
MeSH Terms: conditions — Abortion, Habitual; Infertility; Anemia, Iron-Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples taken as part of routine clinical practice: Total serum iron, serum ferritin, transferrin, transferrin saturation, C-reactive protein
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with infertility: The patient suffers from primary or secondary infertility, defined as the inability to conceive despite frequent unprotected sexual intercourse for at least 12 months.
  Interventions: Diagnostic Test: Blood sample
- Women with recurrent miscarriage: The patient suffers from recurrent miscarriage, defined as three or more consecutive miscarriages before the 20th gestation week with the same partner.
  Interventions: Diagnostic Test: Blood sample
- Healthy controls: The woman does neither suffer from infertility/sterility nor from recurrent miscarriage and is also otherwise healthy with regular cycles.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood samples were taken from a peripheral vein as part of clinical routine. Subsequently, the iron status is determined.

SUMMARY:
Multiple studies suggest a link between the iron status and the development of the endometrium. Therefore, a sufficient iron supply seems to relevant for female fertility and reproduction.

To gain further insight on the effects of iron status on female fertility, a prospective study on infertile women und women with recurrent miscarriage will be conducted. In these, the iron status will be evaluated in detail. In addition, a control group of healthy women without infertility will be enrolled.

DETAILED DESCRIPTION:
The high importance of sufficient iron supply for the human body is without doubt. Notably, it has also been suggested that iron was a central resource in female reproduction.

Women are more prone to iron deficiency than men. It has been stated frequently that blood loss during menstruation was the major cause of lower iron levels in women. On average, women lose about 16 mg of iron for the average menstrual period. This is in line with several studies which demonstrated that women who had menorrhagia were at a higher risk of anemia and iron deficiency anemia. However, the link between menstruation-caused blood loss and iron status is less clear. In previous studies, it was found that higher hemoglobin was associated with a thicker endometrium. An improved body condition, as measured by iron status, might allow women to grow a thicker endometrium despite the fact that a thicker endometrium was associated with greater blood loss.

In addition, reproductive hormones are also implicated in iron status and are also responsible for the sexual dimorphism in iron levels in humans. For example, androgens stimulate the formation of red blood cells and are responsible for their higher hemoglobin levels. The role of estrogens is less clear, since studies have been contradicting. However, studies on the relationship between contraceptive pills and iron status may have provided the biggest clue to the effects of estrogen on iron physiology. Hormonal contraceptive use seems to raise iron stores. Notably, recent evidence suggests that estrogen itself, which also includes the estrogen in contraceptive pills, helps increase absorption of iron.

It has been mentioned that the iron status could be linked with fertility. As part of a larger study on iron supplementation and hair loss, the circumstances of seven women who became pregnant during the supplement intervention has been investigated. Despite the small number of women, this study suggests an intriguing link between iron status and ability to conceive. In addition, a larger, 8-year prospective study of 18,555 premenopausal women in the United States found that women who consumed iron supplements had a significantly lower risk of infertility than women who did not consume iron supplements. Together with the above mentioned observation that women with an improved iron status were able to grow a bigger endometrium, it seems reasonable to assume an influence of iron status on female fertility. Hypothetically, this could lead either to infertility/sterility or to recurrent miscarriage. Notably, one recent small study demonstrated no difference in iron levels between women with recurrent miscarriage and controls. Notably, other parameters of the iron status were not assessed. However, epidemiologic data on iron status and female fertility are scarce. Thus, a prospective study on infertile women und women with recurrent miscarriage will be conducted. In these women, the iron status will be evaluated in detail. In addition, a control group of healthy women without infertility will be enrolled.

ELIGIBILITY:
Women with infertility

Inclusion criteria:

* The patient suffers from primary or secondary infertility, defined as the inability to conceive despite frequent unprotected sexual intercourse for at least 12 months.
* The patient has given her written informed consent after detailed information on the study by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna.
* The patient is >18 and <40 years old.

Exclusion criteria:

* Inflammatoric bowel disease, cardiac insufficiency, chronic kidney disease, any malignant diseases.
* Polycystic ovary syndrome.
* There is no "informed consent".

Women with recurrent miscarriage

Inclusion criteria:

* The patient suffers from recurrent miscarriage, defined as three or more consecutive miscarriages before the 20th gestation week with the same partner.
* The patient has given her written informed consent after detailed information on the study by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna.
* The patient is >18 and <40 years old.

Exclusion criteria:

* Inflammatoric bowel disease, cardiac insufficiency, chronic kidney disease, any malignant diseases.
* Polycystic ovary syndrome
* There is no "informed consent".

Healthy controls

Inclusion criteria:

* The woman does neither suffer from infertility/sterility nor from recurrent miscarriage and is also otherwise healthy with regular cycles.
* The patient has given her written informed consent after detailed information on the study by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna.
* The patient is >18 and <40 years old.

Exclusion criteria:

* Inflammatoric bowel disease, cardiac insufficiency, chronic kidney disease, any malignant diseases.
* Polycystic ovary syndrome
* There is no "informed consent".

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women will be invited to participate by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna, Clinical Division of Gynecologic Endocrinology and Reproductive Medicine, using the above-mentioned criteria in the course of their admission to the outpatient clinics. Potential participants are informed about the procedure, clinical relevance and the balance of risk and benefits incurred through study participation. Patients willing to participate will express this through written affirmation (a "consent form"). Healthy controls will not receive compensation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin in µg/L | 6 months
  Evaluation of a complete iron status including serum ferritin in women with infertility, recurrent miscarriage and healthy controls

SECONDARY OUTCOMES:
serum iron in µg/dL | 6 months
  Evaluation of a complete iron status including serum iron in women with infertility, recurrent miscarriage and healthy controls
transferrin in mg/dL | 6 months
  Evaluation of a complete iron status including transferrin in women with infertility, recurrent miscarriage and healthy controls
transferin-saturation in % | 6 months
  Evaluation of a complete iron status including transferin-saturation in women with infertility, recurrent miscarriage and healthy controls
C-reactive protein mg/dL | 6 months
  Evaluation of a complete iron status including C-reactive protein in women with infertility, recurrent miscarriage and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ott, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller EM. The reproductive ecology of iron in women. Am J Phys Anthropol. 2016 Jan;159(Suppl 61):S172-95. doi: 10.1002/ajpa.22907. PMID 26808104
- [Background] Cook JD. Adaptation in iron metabolism. Am J Clin Nutr. 1990 Feb;51(2):301-8. doi: 10.1093/ajcn/51.2.301. PMID 2407101
- [Background] Hallberg L, Hogdahl AM, Nilsson L, Rybo G. Menstrual blood loss--a population study. Variation at different ages and attempts to define normality. Acta Obstet Gynecol Scand. 1966;45(3):320-51. doi: 10.3109/00016346609158455. No abstract available. PMID 5922481
- [Background] Gao J, Zeng S, Sun BL, Fan HM, Han LH. Menstrual blood loss and hematologic indices in healthy Chinese women. J Reprod Med. 1987 Nov;32(11):822-6. PMID 3430490
- [Background] Cheong RL, Kuizon MD, Tajaon RT. Menstrual blood loss and iron nutrition in Filipino women. Southeast Asian J Trop Med Public Health. 1991 Dec;22(4):595-604. PMID 1820649
- [Background] Clancy KB, Nenko I, Jasienska G. Menstruation does not cause anemia: endometrial thickness correlates positively with erythrocyte count and hemoglobin concentration in premenopausal women. Am J Hum Biol. 2006 Sep-Oct;18(5):710-3. doi: 10.1002/ajhb.20538. PMID 16917885
- [Background] Shahidi NT. Androgens and erythropoiesis. N Engl J Med. 1973 Jul 12;289(2):72-80. doi: 10.1056/NEJM197307122890205. No abstract available. PMID 4575719
- [Background] Yang Q, Jian J, Katz S, Abramson SB, Huang X. 17beta-Estradiol inhibits iron hormone hepcidin through an estrogen responsive element half-site. Endocrinology. 2012 Jul;153(7):3170-8. doi: 10.1210/en.2011-2045. Epub 2012 Apr 25. PMID 22535765
- [Background] Ikeda Y, Tajima S, Izawa-Ishizawa Y, Kihira Y, Ishizawa K, Tomita S, Tsuchiya K, Tamaki T. Estrogen regulates hepcidin expression via GPR30-BMP6-dependent signaling in hepatocytes. PLoS One. 2012;7(7):e40465. doi: 10.1371/journal.pone.0040465. Epub 2012 Jul 11. PMID 22792339
- [Background] Milman N, Kirchhoff M, Jorgensen T. Iron status markers, serum ferritin and hemoglobin in 1359 Danish women in relation to menstruation, hormonal contraception, parity, and postmenopausal hormone treatment. Ann Hematol. 1992 Aug;65(2):96-102. doi: 10.1007/BF01698138. PMID 1511065
- [Background] Milman N, Rosdahl N, Lyhne N, Jorgensen T, Graudal N. Iron status in Danish women aged 35-65 years. Relation to menstruation and method of contraception. Acta Obstet Gynecol Scand. 1993 Nov;72(8):601-5. doi: 10.3109/00016349309021150. PMID 8259744
- [Background] Rushton DH, Ramsay ID, Gilkes JJ, Norris MJ. Ferritin and fertility. Lancet. 1991 Jun 22;337(8756):1554. doi: 10.1016/0140-6736(91)93255-8. No abstract available. PMID 1675411
- [Background] Chavarro JE, Rich-Edwards JW, Rosner BA, Willett WC. Iron intake and risk of ovulatory infertility. Obstet Gynecol. 2006 Nov;108(5):1145-52. doi: 10.1097/01.AOG.0000238333.37423.ab. PMID 17077236
- [Background] Sami AS, Suat E, Alkis I, Karakus Y, Guler S. The role of trace element, mineral, vitamin and total antioxidant status in women with habitual abortion. J Matern Fetal Neonatal Med. 2021 Apr;34(7):1055-1062. doi: 10.1080/14767058.2019.1623872. Epub 2019 Jul 7. PMID 31282231
- [Background] Hou Y, Zhang S, Wang L, Li J, Qu G, He J, Rong H, Ji H, Liu S. Estrogen regulates iron homeostasis through governing hepatic hepcidin expression via an estrogen response element. Gene. 2012 Dec 15;511(2):398-403. doi: 10.1016/j.gene.2012.09.060. Epub 2012 Oct 3. PMID 23041085